CLINICAL TRIAL: NCT02158221
Title: PACAP Induced Migraine Attacks in Patients With High and Low Genetic Load
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Danish Headache Center (Other)
Responsible Party: Principal Investigator, Song Guo, MD, Danish Headache Center
Allocation: Non-Randomized | Model: Parallel | Masking: Double
Other Study IDs: H-2-2013-043
Record Dates: First submitted 2014-06-05; First posted 2014-06-06 (Estimated); Last update posted 2015-02-10 (Estimated); Status verified 2015-02

CONDITIONS: Migraine Without Aura
MeSH Terms: conditions — Migraine without Aura | interventions — Pituitary Adenylate Cyclase-Activating Polypeptide

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor

ARMS (2):
- Migraine patients with high genetic load (Active Comparator): PACAP intravenous infusion 1.5 microgram/min for 20 min
  Interventions: Drug: PACAP
- Migraine patients with low genetic load (Active Comparator): PACAP intravenous infusion 1.5 microgram/min for 20 min
  Interventions: Drug: PACAP

INTERVENTIONS:
Drug: PACAP — Pituitary adenylate cyclase-activating polypeptide (PACAP)
  Other Names: Pituitary adenylate cyclase-activating polypeptide

SUMMARY:
The investigators hypothesized that migraine without patients with many genetic loci associated with migraine (high genetic load) would be more sensitive and get provoked more migraine attacks by PACAP compared to patients with few genetic loci associated with migraine (low genetic load).

DETAILED DESCRIPTION:
Migraine is a very prevalent neurological disorder with a strong genetic factor. The common forms of migraine have a multifactorial and polygenic pattern of inheritance and genetics research is crucial for a deeper understanding of migraine mechanisms. Recently, 12 genetic loci have been identified to be associated with migraine with (MA) and without aura (MA) in four large genome-wide association studies (GWAS). The functional consequences of this genetic variant in humans are yet unknown.

PACAP is a neuropeptide which plays a crucial role in the pathophysiology of migraine and is present in migraine relevant structures. PACAP can induce migraine attacks in MO patients via an adenosine monophosphate (cAMP) dependent pathway. Also, a recent study has showed that intracellular accumulation of cAMP is crucial for the induction of migraine attacks.

The phenotype of the migraine inducing effects of PACAP might therefore be linked to some of the 12 genetic susceptibility loci that have been identified.

ELIGIBILITY:
Inclusion Criteria:

* Migraine without aura patients genotyped for the 12 newly idetified gene variants associated with migraine.

Exclusion Criteria:

* Other primary headache
* A history of cerebrovascular disease and other CNS- disease
* A history suggesting ischaemic heart disease
* Serious somatic and mental disease
* Hypo- or hypertension
* Abuse of alcohol or medicine (opioid analgesics).
* Pregnant or breastfeeding women.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 32 (Actual)
Dates: Start 2014-06; Primary Completion 2014-11 (Actual); Study Completion 2014-12 (Actual)

PRIMARY OUTCOMES:
Incidence of migraine attacks induced by PACAP in patients with high and low genetic load. | Change from baseline in headache intensity at 12 hours after the start of infusion of PACAP
  The difference in incidence of migraine-like attacks after PACAP between patients with and without high genetic load and patients with low genetic load using verbal rating scale (VRS).

SECONDARY OUTCOMES:
Incidence of headache induced by PACAP in patients with high and low genetic load. | Change from baseline in headache intensity at 12 hours after the start of infusion of PACAP
  The difference in area under the curve (AUC) for headache intensity scores (0-12 hours) after infusion of PACAP

CONTACTS AND LOCATIONS:
Locations (1):
- Danish Headache Center & Department of Neurology, Copenhagen, Glostrup, Denmark